CLINICAL TRIAL: NCT07002827
Title: Effect of Single vs Repeated Cycles of a Combination of Granulocyte Colony Stimulating Factor and Darbepoetin vs Standard Medical Treatment on Immunometabolic Profile in Patient With Early Decompensated Cirrhosis -A Pilot Randomised Controlled Trial.
Brief Title: Effect of Single vs Repeated Cycles of a Combination of Granulocyte Colony Stimulating Factor and Darbepoetin vs Standard Medical Treatment on Immunometabolic Profile in Patient With Early Decompensated Cirrhosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-73
Record Dates: First submitted 2025-05-03; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Decompensated Liver Cirrhosis
MeSH Terms: interventions — Darbepoetin alfa; Granulocyte Colony-Stimulating Factor; Lactulose; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Medical treatment (Active Comparator): Standard medical therapy including lactulose, bowel enema and albumin will be continued in both groups.
  Interventions: Drug: Lactulose; Biological: Albumin
- Single cycle of G-CSF + darbepoetin and standard medical treatment (Experimental): * G-CSF will be given at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30.
  * Darbepoetin will be given s/c at dose of 40 mcg once a week (total 4 doses) for 1 month.
  * Standard medical therapy including lactulose, bowel enema and albumin will be continued in both groups.
  Interventions: Drug: Darbepoetin; Drug: G-CSF; Drug: Lactulose; Biological: Albumin
- Three cycles of G-CSF + darbepoetin and standard medical treatment (1-month, 3-month, and 5-month) (Experimental): * G-CSF will be given at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30.
  * Darbepoetin will be given s/c at dose of 40 mcg once a week (total 4 doses) for 1 month.
  * Standard medical therapy including lactulose, bowel enema and albumin will be continued in both groups.
  Interventions: Drug: Darbepoetin; Drug: G-CSF; Drug: Lactulose; Biological: Albumin

INTERVENTIONS:
Drug: Darbepoetin — Darbepoetin will be given s/c at dose of 40 mcg once a week (total 4 doses) for 1 month
  Arms: Single cycle of G-CSF + darbepoetin and standard medical treatment; Three cycles of G-CSF + darbepoetin and standard medical treatment (1-month, 3-month, and 5-month)
Drug: G-CSF — G-CSF will be given at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30
  Arms: Single cycle of G-CSF + darbepoetin and standard medical treatment; Three cycles of G-CSF + darbepoetin and standard medical treatment (1-month, 3-month, and 5-month)
Drug: Lactulose — Standard Medical Tretament part
Biological: Albumin — Standard Medical Tretament part

SUMMARY:
Exogenous growth factor-mobilized bone marrow (BM) stem cells(G-CSF) and DARBEPOETIN use have shown a differential response in the management of decompensated cirrhosis (DC) with improved survival, CTP and MELD scores. This study was designed to evaluate potential clinical benefit of repeated cycles of granulocyte-colony stimulating factor (G-CSF) and DARBEPOETIN versus single cycle on delta change in immunometabolic profile of patients at 6 months assessed in terms of -Change in innate immunity -Monocyte, neutrophils -distribution , function and bioenergetic adaptation .

DETAILED DESCRIPTION:
Aim: To study the efficacy of single vs repeated cycle of Granulocyte Colony Stimulating Factor+ darbopoetin vs standard medical treatmenton immunometabolic profile in patient with early decompensated cirrhosis

Study population:

* Age 18-70 years
* Early decompensated cirrhosis MELD < 16 , CTP < 9B
* Uncomplicated ascites
* A Prospective Randomized Controlled Trial.
* Single Centre.
* Open label.
* Block Randomization will be done , it will be implemented by IWRS method.
* The study will be conducted in Department of Hepatology, ILBS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Decompensated cirrhosis patients
3. Uncomplicated ascites,
4. CTP ≤ 9B and MELD <16
5. BM Hematopoietic stem cell reserve > 0.4
6. Given informed consent

Exclusion Criteria:

1. Patients with age less than 18 years or more than 65 years
2. Lack of informed consent
3. Patients with a history of serious allergic reactions to the active component, filgrastim, other human granulocyte colony-stimulating factors, or any of the ingredients
4. Evidence of alcoholic hepatitis/active alcohol abuse last intake ≤ 3 months
5. Suspected autoimmune hepatitis (ANA/ASMA-positive in titers 1:80 and/ or IgG 1.5 times upper limit of normal),
6. Hemolytic anaemia -Sickle cell disease or thalassemia
7. Patients with Grade III ascites /complicated ascites
8. Patients with large spleen (size ≥ 15cm)
9. Recent variceal bleeding in less than 42 days
10. Patients with any focus of sepsis as proven by culture positivity or presence of spontaneous Bacterial Peritonitis (SBP)
11. H/o Seizures
12. Hepatocellular Carcinoma (HCC) or other malignancy
13. Acute Kidney Injury (AKI) with serum Creatinine >1.5 mg/ dl,
14. Multi-organ failure,
15. Hepatic Encephalopathy or prior history of HE in less than 6months
16. HIV seropositivity,
17. Uncontrolled essential hypertension, CAD /Stroke
18. Massive hydrothorax
19. Pregnancy
20. Viral etiology of liver disease
21. Chronic kidney disease
22. Portal vein thrombosis
23. Planned for LT
24. Bone marrow hematopoietic stem cells < 0.4

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in innate immunity between the groups. | 6 months
  Innate immunity -Monocyte, neutrophils -distribution , function and bioenergetic adaptation

SECONDARY OUTCOMES:
Proportion of participants developed new-onset of LRE (such as ascites, HE, AKI, bleed and sepsis) or show mortality in all the groups. | 6 months
Cumulative incidence of second decompensation in all the groups. | 6 months & 1 year
Transplant-free survival. | 6 months & 1 year
Number of participants with improvement in liver disease severity indices (CTP). | 6 months
Number of participants with improvement in liver disease severity indices (MELD). | 6 months
Number of participants with change in adaptive immunity(T-cell, B-cell and NK cells distribution only ) | 6 months
Number of participants with change in inflammation (a panel of pro and anti-inflammatory cytokines). | 6 months
Change in gcsf levels and EPO levels at baseline and completion of each cycle. | 6 months
Proportion of participants completing treatment without major adverse effects; | 6 months
Number of participants with change in peripheral blood CD34+ Hematopoietic Stem Cells count at 6months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Manoj Kumar Sharma, DM, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided